CLINICAL TRIAL: NCT06452498
Title: Metformin for the Prolongation of Pregnancy in Preterm Preeclampsia
Brief Title: Preeclampsia Intervention Netherlands
Acronym: PI-NL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amsterdam UMC (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Dr Rebecca C. Painter, Prof. dr., Amsterdam UMC
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PI-NL trial; 2023-510382-10-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-31; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pre-Eclampsia Onset Less Than 37 Weeks; Pre-Eclampsia; Pre-Eclampsia; Complicating Pregnancy; Pre-Eclampsia as Antepartum Condition; Pre-eclampsia or Eclampsia With Pre-existing Hypertension; Pre-Eclampsia; Affecting Fetus; HELLP Syndrome Complicating Pregnancy; HELLP Syndrome; HELLP
Keywords: Preterm Preeclampsia; Metformin; RCT; Placebo; Gestational Prolongation; Treatment; Pregnancy; Multicenter; Preterm; HELLP Syndrome; Hypertensive disorders of pregnancy; Preeclampsia; Randomized controlled trial
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications; HELLP Syndrome; Premature Birth | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Two-arm trial with intervention arm (metformin) and comparator arm (placebo), aside from usual care for all patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, treating clinicians, and trial investigators will be blinded to the allocated treatment. Masking will be removed once the database has been locked, after which data analysis will be undertaken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Metformin 3000 mg divided by three daily doses (3 times 2 capsules of 500 mg; following a step-up schedule) from randomization till delivery, aside from usual preterm preeclampsia care.
  Interventions: Drug: Metformin Hydrochloride
- Placebo (Placebo Comparator): Placebo, divided by three daily doses (3 times 2 capsules; following a step-up schedule) from randomization till delivery, aside from usual preterm preeclampsia care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin Hydrochloride encapsulated immediate-release tablet of 500 mg, backfilled with cellulose.
  Other Names: Metformin; Metformin HCl
  Arms: Metformin
Drug: Placebo — Capsule filled with cellulose.
  Arms: Placebo

SUMMARY:
The goal of this study is to find out if pregnant individuals with preterm preeclampsia (PE) who are treated with metformin can stay pregnant for longer, and if this is safe(r) for the mother and child. Preterm PE affects about 1 in 100 pregnant individuals in the Netherlands. Signs of preterm PE can be high blood pressure and protein in the urine in the second half of pregnancy (but before 32-34 weeks of pregnancy). Other symptoms can develop, such as problems with blood clotting and how well the blood cells, liver, lungs, and brain work. The disease can lead to serious complications for both the mother and child. The only way to cure preterm PE is to make sure the child is born, and many times, children have to be delivered (very) early (before 37 weeks). Children born (very) early can suffer from infections, breathing difficulties, and problems in their development.

Metformin is a medicine used to treat high blood sugar during and outside of pregnancy. In a previous study in South Africa, women with preterm PE that used metformin were able to safely remain pregnant for an extra week. Similarly, the main goal of the Preeclampsia Intervention NetherLands (PI-NL) study is to see if patients with preterm PE in the Netherlands that use metformin can remain pregnant for a longer time than patients taking a placebo. A placebo is a look-a-like capsule that contains no active ingredients. Researchers, the treating medical team, and participants will not know which participant gets which treatment. In addition, all participants will receive the standard care that all preterm PE patients get.

DETAILED DESCRIPTION:
Preterm preeclampsia (PE) is a severe hypertensive disorder of pregnancy and a major cause of maternal and perinatal morbidity and mortality. Currently, the only treatment to halt disease progression is delivery of the dysfunctional placenta and thereby the child. This often happens prematurely. Being able to safely (for mother and child) extend pregnancy, even by a few days, is expected to reduce the short- and long-term risks associated with (severe) prematurity. Preclinical and recent clinical evidence presents metformin, a drug commonly used to treat diabetes in and outside of pregnancy, as a promising treatment candidate for preterm PE. Metformin might reduce inflammation, oxidative stress, and anti-angiogenesis, and improve endothelial function. In a recent South African trial, use of metformin was associated with a safe median 7.6 day prolongation of pregnancy in women with preterm PE, compared to placebo. There was a nonsignificant increase in the neonatal birthweight and a decrease in the length of stay in any neonatal nursery. Metformin did not lead to any serious adverse events.

The goal of this multicenter, triple-blind, randomized placebo-controlled trial is to investigate whether metformin can safely prolong gestation in patients with preterm PE in the Dutch population. Secondary outcomes include composite adverse maternal, fetal, and neonatal outcomes. Cost-effectiveness of the treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria

All of the following:

* Aged 18 years or older
* Singleton pregnancy
* Gestational age between 23+0 and 31+6 weeks
* A diagnosis of preterm preeclampsia, defined according to modified International Society for the Study of Hypertension in Pregnancy (ISSHP) classification, including only those who have proteinuria (≥300 mg of protein in a 24-hour urine specimen or a protein-creatinine-ratio >50 in a single urine sample)
* Estimated fetal weight >400 grams
* No clear indication (maternal or fetal) or intention, by both the treating multidisciplinary team and the patient after counseling, to immediately deliver (or directly after corticosteroid administration) or to terminate the pregnancy otherwise.
* Ability to understand English or Dutch
* Ability and willingness to provide written informed consent

Exclusion Criteria

Any of the following:

* Current use of metformin or a clinical indication for the use of metformin
* A decision for immediate delivery (including cases where corticosteroids are administered with planned delivery directly after completion of treatment) or termination of pregnancy (e.g., due to disease severity in the patient combined with a dismal prognosis for the fetus), as made by the treating multidisciplinary team and the parent(s)
* Contraindication(s) for the use of metformin (e.g., severe renal insufficiency, acute metabolic acidosis, severe liver insufficiency)
* Use of drugs that might interact with metformin
* Suspicion of a major fetal anomaly and/or chromosomal abnormality
* Unable or unwilling to (completely) understand or provide informed consent, due to language, culture, or other barriers

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of days between randomization and delivery | Time between randomization and delivery (up to 37 weeks of gestation)
  Prolongation of gestation

SECONDARY OUTCOMES:
Number of participants reaching a composite maternal adverse outcome | Randomization till 90 days postpartum (unless otherwise specified)
  Combined endpoint of maternal death (during pregnancy or within 42 days postpartum), eclampsia, pulmonary edema, severe renal impairment, cerebrovascular accident, placental abruption, and/or liver hematoma or rupture.
Number of participants reaching a composite fetal adverse outcome | Randomization till delivery (up to 37 weeks of gestation)
  Combined endpoint of intrauterine fetal demise, suboptimal fetal condition based on CTG, and fetal growth restriction.
Number of participants reaching a composite neonatal adverse outcome | Birth till 90 days after birth (unless otherwise specified)
  Combined endpoint of neonatal death (within 28 days after birth), grade 3 or 4 intraventricular hemorrhage, retinopathy of prematurity requiring treatment, necrotizing enterocolitis (grade II or higher), bronchopulmonary dysplasia, neonatal sepsis, and cystic periventricular leukomalacia (grade II or higher)

OTHER OUTCOMES:
Maternal individual exploratory outcomes | Randomization till 90 days postpartum (unless otherwise specified)
  Number of participants experiencing each of the following: maternal death, cerebrovascular event, eclampsia, cortical blindness, pulmonary edema, AKI, liver hematoma/rupture, placental abruption, retinal detachment, postpartum hemorrhage, HELLP syndrome, severe elevated liver enzymes, low platelets, left ventricular heart failure, PRES, DIC, thromboembolic disease, need for dialysis due to renal failure, admission to high or ICU, need for intubation and mechanical ventilation
Fetal individual exploratory outcomes | Randomization till 90 days postpartum (unless otherwise specified)
  Number of participants experiencing each of the following: intrauterine or intrapartum fetal death, reversed end diastolic flow in umbilical artery on at least 2 occasions, redistribution in the middle cerebral artery, absent or reversed a-wave in ductus venosus, suboptimal fetal condition based on CTG.
Neonatal individual exploratory outcomes | Randomization till 90 days postpartum (unless otherwise specified)
  Number of participants experiencing each of the following: neonatal death within 28 days after birth, neonatal death between 29 and 90 days after birth, growth restriction at birth, Apgar score < 7 at 5 min, umbilical artery pH < 7.10, neonatal hypoglycemia, neonatal seizures, intraventricular hemorrhage, necrotizing enterocolitis, retinopathy of the premature, pulmonary insufficiency of the preterm infant, bronchopulmonary dysplasia, cystic periventricular leukomalacia, patent ductus arteriosus, persistent pulmonary hypertension, surfactant use within 72 hours after birth, need for respiratory support, admission to NICU.
Mean neonatal birthweight | Within the first 24 hours after birth
  In grams
Median neonatal length of stay in any neonatal nursery, including NICU | Birth till 90 days postpartum
  In days
Incremental cost-effectiveness ratios (ICERs; exploratory) | Start of pregnancy till 90 days postpartum
  Determined through length of maternal stay in hospital (and specifically ICU), neonatal length of stay in hospital (and specifically NICU), other health care utilization (based on iMCQ questionnaire, maternal and neonatal use of medication during pregnancy and after birth), loss of productivity (measured with iPCQ questionnaire), quality-of-life (score on EQ-5D-5L).
Rate of diarrhea, nausea/vomiting, abdominal pain, headache (all based on PHASE-20 questionnaire), lactic acidosis, and hypoglycemia (individually) | Randomization till delivery (up to 37 weeks of gestation)
  Tolerability and safety of metformin
Score on PROMIS Anxiety 8a Short Form | Randomization till 90 days postpartum
  Maternal anxiety
Score on EPDS | Randomization till 90 days postpartum
  Maternal depressive symptoms
Score on Rosenberg Self-Esteem Scale | Randomization till 90 days postpartum
  Maternal self-esteem
Score on City Birth Trauma Scale | Randomization till 90 days postpartum
  Child-related PTSD

CONTACTS AND LOCATIONS:
Overall Officials: R.C. Painter, Prof, MD, PhD, Principal Investigator — Amsterdam UMC

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to collaborate with researchers doing similar Preeclampsia Intervention (PI) trials.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code